CLINICAL TRIAL: NCT00087568
Title: An Open-label, Multicenter, Efficacy and Safety Study of Pegasys® Plus Ribavirin in Patients With Chronic HCV Infection Who Are Unable to Tolerate or Who Do Not Respond to 12 Weeks of Therapy With PEGIntron ® Plus Ribavirin
Brief Title: A Study of PEGASYS (Peginterferon Alfa-2a (40KD)) in Combination With Ribavirin in Patients With Chronic Hepatitis C (CHC) Previously Treated With PEG-Intron + Ribavirin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML16965
Record Dates: First submitted 2004-07-12; First posted 2004-07-14 (Estimated); Results first posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-05

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a

ARMS (2):
- Non-Responders (Experimental): Participants will receive Pegasys 180 micro grams (µg or mcg) subcutaneously (SC) once a week and ribavirin 1000 or 1200 milligrams per day [(mg/day), < or >=75 kilogram (Kg) body weight, respectively], orally in divided doses for 60 weeks.
  Interventions: Drug: Ribavirin; Drug: peginterferon alfa-2a [Pegasys]
- Non-Tolerators (Experimental): Participants will receive Pegasys 180 µg subcutaneously (SC) once a week and ribavirin 1000 or 1200 mg/day (< or >=75 kg body weight, respectively) orally in divided doses for 36 weeks.
  Interventions: Drug: Ribavirin; Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: Ribavirin — 1000/1200mg po bid for 36 or 60 weeks
Drug: peginterferon alfa-2a [Pegasys] — 180 micrograms weekly for 36 weeks (non-responders) or 60 weeks (non-tolerators)

SUMMARY:
This study will evaluate the efficacy, safety and tolerability of PEGASYS plus ribavirin in patients with CHC who could not tolerate or were not responsive to 12 weeks of therapy with PEG-Intron plus ribavirin. The anticipated time on study treatment is 1-2 years, and the target sample size is >100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients at least 18 years of age
* CHC infection, genotype 1
* unable to tolerate or not responsive to PEG-Intron + ribavirin therapy after 12 weeks of treatment
* use of 2 forms of contraception during the study in both men and women

Exclusion Criteria:

* women who are pregnant or breast-feeding
* medical condition associated with chronic liver disease (eg, hemochromatosis, autoimmune hepatitis, alcoholic liver disease, toxin exposures)
* patients with decompensated cirrhosis
* patients receiving any systemic antiviral therapy or investigational drug, other than PEG-Intron + ribavirin, 24 weeks prior to the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2003-01; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- United States (25):
  - Bakersfield, California
  - Pasadena, California
  - San Diego, California
  - San Mateo, California
  - Bradenton, Florida
  - Miami, Florida
  - Orlando, Florida
  - Austell, Georgia
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Kansas City, Missouri
  - Bayside, New York
  - Brooklyn, New York
  - Manhasset, New York
  - New York, New York
  - Valhalla, New York
  - Statesville, North Carolina
  - Cincinnati, Ohio
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Houston, Texas
  - Fairfax, Virginia
  - Richmond, Virginia
  - Tacoma, Washington

REFERENCES:
- [Derived] Bonkovsky HL, Tice AD, Yapp RG, Bodenheimer HC Jr, Monto A, Rossi SJ, Sulkowski MS. Efficacy and safety of peginterferon alfa-2a/ribavirin in methadone maintenance patients: randomized comparison of direct observed therapy and self-administration. Am J Gastroenterol. 2008 Nov;103(11):2757-65. doi: 10.1111/j.1572-0241.2008.02065.x. Epub 2008 Aug 5. PMID 18684176
- [Derived] Rustgi VK, Esposito S, Hamzeh FM, Shiffman ML. Peginterferon alfa-2a/ribavirin in hepatitis C virus patients nontolerant or nonresponsive to peginterferon alfa-2b/ribavirin. Aliment Pharmacol Ther. 2008 Mar 1;27(5):433-40. doi: 10.1111/j.1365-2036.2007.03587.x. Epub 2007 Dec 10. PMID 18081737

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 29 Jan 2003 to 24 Mar 2006 across 14 centers in the United States.
Pre-assignment Details: A total of 80 participants (40 non-tolerators and 40 non-responders) were planned; however, 57 participants were enrolled only after receiving 12 weeks of PEG-Intron plus ribavirin therapy and received the study medication (25 non-tolerators and 32 non-responders).
Groups:
- Non-Responders: Participants received Pegasys 180 micrograms (µg) subcutaneously (SC) once a week and ribavirin 1000 or 1200 milligrams per day [mg/day (< or >=75 kg body weight, respectively)], orally in divided doses for 60 weeks.
- Non-Tolerators: Participants received Pegasys 180 µg subcutaneously (SC) once a week and ribavirin 1000 or 1200 mg/day (< or >=75 kg body weight, respectively) orally in divided doses for 36 weeks.
Period: Overall Study
Arm/Group | Non-Responders | Non-Tolerators
Started | 32 | 25
Completed | 2 | 23
Not Completed | 30 | 2
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lack of Efficacy | 24 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all enrolled participants who received at least one dose of study medication (Pegasys or ribavirin).
Groups:
- Non-Responders: Participants received Pegasys 180 µg subcutaneously (SC) once a week and ribavirin 1000 or 1200 mg/day (< or >=75 kg body weight, respectively), orally in divided doses for 60 weeks.
- Total: Total of all reporting groups
Arm/Group | Non-Responders | Non-Tolerators | Total
Number analyzed (Participants) | 32 | 25 | 57
Age, Continuous [Median (Full Range); unit: years] | 47.0 [32 to 68] | 49.0 [35 to 66] | 49.0 [32 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 22
  Male | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Pegasys and Ribavirin Therapy Completers
Description: Therapy completers were defined as all participants who had demonstrable viremia after 12 weeks of Pegasys plus ribavirin therapy (who were to be discontinued for lack of efficacy), non-tolerators who completed 36 weeks of Pegasys plus ribavirin therapy, and non-responders who completed 60 weeks of Pegasys plus ribavirin therapy. Study completers included all participants who completed the planned treatment period (36 weeks for non-tolerators and 60 weeks for non-responders) and the 24-week treatment-free follow-up period and participants in either group who were prematurely discontinued per protocol due to insufficient therapeutic response at Week 12.
Time Frame: 36 weeks for Non-Tolerators and 60 weeks for Non-Responders
Population: Safety Population included all enrolled participants who received at least one dose of study medication (Pegasys or ribavirin) and had at least one post-baseline safety assessment which defined as clinical adverse event, laboratory or vital sign data, physical examination finding, Beck Depression Inventory (BDI-II), or Fatigue severity score (FSS).
Measure: Number; unit: Participants
Arm/Group | Non-Responders | Non-Tolerators
Number analyzed (Participants) | 32 | 25
Participants
  Completing 36 weeks | 3 | 23
  Completing 60 weeks | 2 | 23

2. Secondary Outcome: Number of Participants With >=2-log10 Decrease or Undetectable (<60 International Units Per Milliliter) Hepatitis C Virus-ribonucleic Acid Over Time
Description: Sustained virological response (SVR) is defined as undetectable Hepatitis C virus-ribonucleic acid (HCV RNA)(<60 International units per milliliter) or HCV RNA for >=2-log10 decrease in viral titre, 24 weeks after the end of treatment. A participant was classified as non-responder (SVR not achieved) if HCV RNA was detectable at the completion of antiviral treatment, at Week 24 post or at any time between Week 24 and completion of antiviral treatment. HCV RNA measured prior to or on the date of the first dose of Pegasys plus ribavirin was used as the baseline in all HCV RNA analyses.
Time Frame: Weeks 4, 12, 24, 36, 48, 60, and 84
Population: Intent to treat (ITT) Population included all enrolled participants who received at least one dose of study medication (Pegasys or ribavirin).
Measure: Number; unit: Participants
Arm/Group | Non-Responders | Non-Tolerators
Number analyzed (Participants) | 32 | 25
Participants
  Week 4 | 1 | 16
  Week 12 | 4 | 24
  Week 24 | 1 | 21
  Week 36 | 2 | 21
  Week 48 | 1 | 11
  Week 60 | 2 | 14
  Week 84 | 1 | 0

3. Secondary Outcome: Number of Participants With Normal Serum Alanine Transaminase Levels Over Time
Description: The number of participants with serum alanine transaminase (ALT) concentration within the normal range at each time point assessed. Upper limit of normal serum ALT for men is 43 International units per liter (IU/L) and for women is 34 IU/L.
Time Frame: Baseline (Week 0), Weeks 4, 12, 24, 36, 48, 60, and 84
Population: ITT Population included all enrolled participants who received at least one dose of study medication (Pegasys or ribavirin).
Measure: Number; unit: Participants
Arm/Group | Non-Responders | Non-Tolerators
Number analyzed (Participants) | 32 | 25
Participants
  Baseline | 21 | 21
  Week 4 | 18 | 19
  Week 12 | 9 | 19
  Week 24 | 6 | 16
  Week 36 | 3 | 15
  Week 48 | 3 | 14
  Week 60 | 1 | 15
  Week 84 | 1 | 0

4. Secondary Outcome: Number of Participants With Serious Adverse Events and Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An adverse event could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Pre-existing conditions that worsened during the study were also to be reported as adverse events. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is medically significant or requires intervention to prevent one or other of the outcomes listed above.
Time Frame: Up to Week 84
Population: Safety Population included all enrolled participants who received at least one dose of study medication (Pegasys or ribavirin) and had at least one post-baseline safety assessment (defined as clinical adverse event, laboratory or vital sign data, physical examination finding, BDI-II score, or FSS score).
Measure: Number; unit: Participants
Arm/Group | Non-Responders | Non-Tolerators
Number analyzed (Participants) | 32 | 25
Participants
  any SAE | 1 | 1
  any AE | 29 | 23

5. Secondary Outcome: Mean Score of Beck Depression Inventory Over Time
Description: The Beck Depression Inventory (BDI-II) is a questionnaire with groups of statements in which the patient is asked to select the statement that most clearly describes the way he/she has felt in the past two weeks, including today. The score for each group is tallied and the ranges of scores are used as guidelines for measuring the degree of depression. For this study, scores are defined as follows: 0 to 15 as minimal, 16 to 21 as mild, 22 to 30 as moderate, and 31 to 63 as severe. The questionnaire was in two areas (changes in sleeping pattern and changes in appetite), selections 1, 2, and 3 contained options for both more and less with respect to the area of interest. Four statements (labelled 0, 1, 2, and 3) were offered that described the area of interest, with 0 indicating no effect and 3 indicating the worst effect. The individual area scores were summed to provide a total score.
Time Frame: Baseline (Week 0); Weeks 4, 12, 24, 36, 48, 60, and 84
Population: Safety Population included all enrolled participants who received at least one dose of study drug and had at least one post-baseline safety assessment (a clinical adverse event, laboratory or vital sign data, physical examination finding, BDI-II score, or FSS score). n = number of participants available at the particular time for assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Non-Responders | Non-Tolerators
Number analyzed (Participants) | 32 | 25
Units on a scale
  Baseline, (n = 32, 25) | 10.93 (9.32) | 15.03 (7.56)
  Week 4, (n = 31, 24) | 9.52 (8.34) | 10.68 (5.64)
  Week 12, (n = 27, 24) | 8.63 (7.74) | 10.76 (7.97)
  Week 24, (n = 2, 23) | 3.75 (0.64) | 11.26 (7.30)
  Week 36, (n = 3, 19) | 5.40 (3.83) | 8.65 (5.73)
  Week 48, (n = 2, 21) | 6.15 (4.03) | 4.30 (4.54)
  Week 60, (n = 2, 21) | 3.00 (4.24) | 3.62 (3.40)
  Week 84, (n = 2, 0) | 1.50 (2.12) | NA (NA) — No participants in the "Non-Tolerators" provided data at Week 84

6. Secondary Outcome: Mean Score of Fatigue Severity Over Time
Description: The Fatigue severity score (FSS) scale has a series of questions designed to assess tiredness, lack of energy, or total body give-out. Participants were to react to nine statements regarding fatigue over the previous 2 weeks, each on a scale (1 = completely agree, 7 = completely disagree). The FSS is the average of the scores on the 9 questions; ranging from 1-7, with lower scores indicating less fatigue. In addition, participants were to react to how much fatigue they had in the past 2 or 4 weeks by marking on a visual analogue scale labelled at one end with "no fatigue" ('0' being the best) and at the other end with "greater fatigue" ('100' being the worst). Longer distance on the scale from "no fatigue" indicated "greater fatigue". FSS values are presented based on questionnaire and visual analog scale.
Time Frame: Baseline (Week 0); Weeks 4, 12, 24, 36, 48, 60, and 84
Population: Safety Population included all the enrolled participants who received at least one dose of study medication and had at least one post-baseline safety assessment (a clinical adverse event, laboratory or vital sign data, physical examination finding, or FSS score). n = number of participants available at the particular time for assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Non-Responders | Non-Tolerators
Number analyzed (Participants) | 32 | 25
Units on a scale
  Total FSS, Baseline, (n = 32, 25) | 4.66 (1.73) | 5.14 (1.27)
  Total FSS, Week 4, (n = 31, 24) | 4.27 (1.76) | 4.50 (1.59)
  Total FSS, Week 12, (n = 27, 24) | 4.09 (1.84) | 4.72 (1.72)
  Total FSS, Week 24, (n = 2, 23) | 1.33 (0.47) | 4.99 (1.56)
  Total FSS, Week 36,(n = 3, 19) | 2.52 (1.41) | 4.62 (1.75)
  Total FSS, Week 48, (n = 2, 21) | 2.22 (1.73) | 3.17 (1.17)
  Total FSS, Week 60, (n = 2, 20) | 2.44 (2.04) | 2.97 (1.13)
  Total FSS, Week 84, (n = 2, 0) | 1.61 (0.86) | NA (NA) — No participants in the "Non-Tolerators" provided data at Week 84
  Visual analog based FSS, Baseline, (n = 32, 25) | 48.72 (25.64) | 61.92 (23.38)
  Visual analog based FSS, Week 4, (n = 31, 24) | 47.87 (29.67) | 52.08 (25.92)
  Visual analog based FSS, Week 12, (n = 27, 24) | 52.15 (31.52) | 55.00 (26.96)
  Visual analog based FSS, Week 24, (n = 2, 23) | 54.50 (19.09) | 56.52 (28.70)
  Visual analog based FSS, Week 36, (n = 3, 19) | 47.33 (16.65) | 48.79 (29.09)
  Visual analog based FSS, Week 48, (n = 2, 21) | 26.00 (1.41) | 25.24 (22.27)
  Visual analog based FSS, Week 60, (n = 2, 20 | 31.00 (2.83) | 31.55 (32.45)
  Visual analog based FSS, Week 84, (n = 2, 0) | 21.50 (16.26) | NA (NA) — No participants in the "Non-Tolerators" provided data at Week 84

7. Secondary Outcome: Number of Participants With Individual Flu-like Symptom
Description: Participants were asked to complete a flu-like symptom questionnaire at screening, study baseline, and at all subsequent scheduled visits. The "yes/no" questionnaire evaluated the incidence of headache, fever, myalgia, and chills. If a participant answered "yes" to the question "Has the patient experienced any flu-like symptoms since the last visit?" all among headache, fever, muscle aches (myalgia), and chills that applied were to be marked. If any of the experienced symptoms was newly reported or had worsened, a corresponding adverse event was to be reported.
Time Frame: Baseline (Week 0); Weeks 12, 36, 60 and 84
Population: Safety Population included all the enrolled participants who received at least one dose of study medication and had at least one post-baseline safety assessment (a clinical adverse event, laboratory or vital sign data, physical examination data, BDI-II score, or FSS score). n = number of participants available at the particular time of assessment.
Measure: Number; unit: Participants
Arm/Group | Non-Responders | Non-Tolerators
Number analyzed (Participants) | 32 | 25
Participants
  Baseline, Headache, (n = 32, 25) | 16 | 19
  Baseline, Fever, (n = 32, 25) | 10 | 14
  Baseline, Muscle aches, (n = 32, 25) | 17 | 21
  Baseline, Chills, (n = 32, 25) | 12 | 17
  Week 12, Headache, (n = 27, 24) | 13 | 13
  Week 12, Fever, (n = 27, 24) | 3 | 5
  Week 12, Muscle aches, (n = 27, 24) | 8 | 10
  Week 12, Chills, (n = 27, 24) | 2 | 5
  Week 36, Headache, (n = 3, 19) | 2 | 10
  Week 36, Fever, (n = 3, 19) | 1 | 3
  Week 36, Muscle aches, (n = 3, 19) | 1 | 8
  Week 36, Chills, (n = 3, 19) | 1 | 7
  Week 60, Headache, (n = 2, 22) | 0 | 1
  Week 60, Fever, (n = 2, 22) | 0 | 0
  Week 60, Muscle aches, (n = 2, 22) | 0 | 2
  Week 60, Chills, (n = 2, 22) | 0 | 1
  Week 84, Headache, (n = 32, 25) | 19 | 18
  Week 84, Fever, (n = 32, 25) | 10 | 14
  Week 84, Muscle aches, (n = 32, 25) | 18 | 19
  Week 84, Chills, (n = 32, 25) | 9 | 15

8. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities
Description: Analysis was performed for hematology, clinical chemistry, thyroid function, and urinalysis. Normal ranges of the parameters were: Haematocrit (fraction): 0.37 - 0.49, Haemoglobin (g/L): 130 - 180 , Platelets (G/L): 150 - 350, White blood cell (G/L): 4.5 - 11.0, Lymphocytes (G/L): 1.00 - 4.80, Neutrophils (G/L): 1.80 - 7.70, Prothrombin Time in Seconds (sec): not defined, Prothrombin Time, normalized (ratio): 0.70 - 1.30, Partial thromboplastin Time (sec): 22.1 - 34.1, Aspartate transaminase (AST) or serum glutamate oxaloacetate transaminase (SGOT) in IU/L: 0 - 40, Alkaline Phosphatase (IU/L): 0 - 115, ALT or serum glutamate pyruvate transaminase (SGPT) in (IU/L): 0-55, Total Bilirubin (umol/L): 0 -17, Thyroxine (T4) (nmol/L): 58 -140, Thyroid-stimulating hormone (TSH, [U/mL]): 0.0 - 5.0, Triglycerides (mmol/L): 0.45 - 1.69, Phosphate (mmol/L): 0.84 - 1.45, Uric Acid (umol/L): 214 - 506
Time Frame: Up to Week 84
Population: Safety Population included all the enrolled participants who received at least one dose of study medication and had at least one post-baseline safety assessment (a clinical adverse event, laboratory, vital sign, or physical examination finding, BDI-II score, or FSS score). 'n' = number of participants available at the time of assessment.
Measure: Number; unit: participants
Arm/Group | Non-Responders | Non-Tolerators
Number analyzed (Participants) | 32 | 25
participants
  Hematocrit (fraction) - Low (n = 32, 25) | 5 | 3
  Hemoglobin-Low (n = 32, 25) | 5 | 6
  Platelets - Low (n = 32, 25) | 6 | 3
  WBC (White blood cells)-High (n = 32, 25) | 1 | 1
  WBC (White blood cells) - Low (n = 32, 25) | 11 | 13
  Lymphocytes - High (n = 32, 25) | 1 | 0
  Lymphocytes - Low (n = 32, 25) | 6 | 5
  Neutrophils - High (n = 32, 25) | 3 | 1
  Neutrophils - Low (n = 32, 25) | 19 | 20
  Partial thromboplastin Time - High (n = 32, 25) | 1 | 1
  Prothrombin time - High (n = 32, 25) | 0 | 1
  SGOT - High (n = 32, 25) | 14 | 8
  SGPT - High (n = 32, 25) | 9 | 9
  Alkaline phosphatase - High (n = 32, 25) | 1 | 0
  Phosphate - High (n = 32, 25) | 1 | 1
  Phosphate - Low (n = 32, 25) | 2 | 3
  Uric acid - High (n = 32, 25) | 1 | 0
  Triglycerides - High (n = 32, 25) | 10 | 9
  Thyroid-T4 - High (n = 32, 25) | 6 | 0
  Thyroid T4 - Low (n = 32, 25) | 2 | 0
  TSH - High (n = 32, 25) | 3 | 1

9. Secondary Outcome: Number of Participants With Abnormal Vital Signs
Description: Abnormal vital signs were defined as
  1. Systolic blood pressure (BP) below 85 mm Hg or above 180 mm Hg with a change from baseline of > 20%
  2. Diastolic BP above 110 mm Hg with a change from baseline of > 20% where systolic and diastolic BP were pressure exerted by blood on the walls of blood vessels during left ventricular systole and diastole respectively.
  3. Pulse rate below 50 beats per minute and above 120 beats per minute, with a change from baseline of > 20%, where pulse represents the palpation of heartbeat
Time Frame: From screening (Day -21 to Day -1) to Week 84
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Non-Responders | Non-Tolerators
Number analyzed (Participants) | 32 | 25
Participants
  Systolic BP high | 1 | 0
  Systolic BP low | 1 | 0
  Pulse-low | 0 | 1

10. Secondary Outcome: Mean Score for Overall Local Injection Site Reaction
Description: Local injection-site reactions were to be given an overall assessment based on pain or discomfort as Grade 0 for no pain or discomfort, Grade 1 for mild tenderness at the injection site, Grade 2 for moderate pain without limitation of usual activities, Grade 3 for severe pain requiring prescription non-topical analgesics or limiting usual activities, Grade 4 for a reaction that resulted in a new hospitalization, prolongation of hospitalization, death, or a persistent or significant disability/incapacity, or was life threatening or medically significant. Adverse events related to the injection site (injection site erythema, hematoma, pain, rash, or reaction) were reported. All of these events were reported as resolved without sequelae.
Time Frame: Baseline (Week 0), Week 4, 12, 24, 36, 48 and 60
Population: Safety Population included all enrolled participants who received at least one dose of study medication and had at least one post-baseline safety assessment (a clinical adverse event, laboratory, vital sign, or physical examination finding, BDI-II score, or FSS score). 'n' = number of participants available at the time of assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Non-Responders | Non-Tolerators
Number analyzed (Participants) | 32 | 25
Units on a scale
  Baseline, (n = 32, 25) | 0.25 (0.57) | 0.48 (0.65)
  Week 4, (n = 31, 24) | 0.03 (0.18) | 0.08 (0.28)
  Week 12, (n = 27, 24) | 0.00 (0.00) | 0.17 (0.38)
  Week 24, (n = 2, 23) | 0.00 (0.00) | 0.09 (0.29)
  Week 36, (n = 3, 19) | 0.00 (0.00) | 0.05 (0.23)
  Week 48, n = (2, 0) | 0.00 (0.00) | NA (NA) — No participants in the "Non-Tolerators" provided data at Week 48 and 60.
  Week 60, n = (2, 0) | 0.00 (0.00) | NA (NA) — No participants in the "Non-Tolerators" provided data at Week 48 and 60.

ADVERSE EVENTS:
Time Frame: Up to Week 84
Description: Safety Population included all the enrolled participants who received at least one dose of study medication (Pegasys or ribavirin) and had at least one post-baseline safety assessment (a clinical adverse event, laboratory, vital sign, or physical examination finding, BDI-II score or FSS score).
Arm/Group | Non-Responders | Non-Tolerators
Serious Adverse Events (participants affected / at risk) | 1/32 | 1/25
Other Adverse Events (participants affected / at risk) | 27/32 | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Responders (N=32) | Non-Tolerators (N=25)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Responders (N=32) | Non-Tolerators (N=25)
FATIGUE (General disorders) | 10 | 7
PYREXIA (General disorders) | 2 | 6
CHILLS (General disorders) | 2 | 3
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 2
INJECTION SITE REACTION (General disorders) | 0 | 3
CHEST DISCOMFORT (General disorders) | 2 | 0
IRRITABILITY (General disorders) | 0 | 2
PAIN (General disorders) | 0 | 2
RASH (Skin and subcutaneous tissue disorders) | 6 | 5
PRURITUS (Skin and subcutaneous tissue disorders) | 3 | 7
ALOPECIA (Skin and subcutaneous tissue disorders) | 5 | 2
HYPOTRICHOSIS (Skin and subcutaneous tissue disorders) | 2 | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 2 | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 3
NAUSEA (Gastrointestinal disorders) | 6 | 4
DIARRHOEA (Gastrointestinal disorders) | 3 | 7
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 0
DRY MOUTH (Gastrointestinal disorders) | 1 | 2
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 2
CONSTIPATION (Gastrointestinal disorders) | 0 | 2
VOMITING (Gastrointestinal disorders) | 0 | 2
INSOMNIA (Psychiatric disorders) | 11 | 6
DEPRESSION (Psychiatric disorders) | 6 | 5
ANXIETY (Psychiatric disorders) | 1 | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 6 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 3
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 2
HEADACHE (Nervous system disorders) | 7 | 5
DIZZINESS (Nervous system disorders) | 1 | 3
HYPOAESTHESIA (Nervous system disorders) | 1 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 2
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 2 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 3
SINUSITIS (Infections and infestations) | 0 | 2
ANAEMIA (Blood and lymphatic system disorders) | 2 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 3 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 2
WEIGHT DECREASED (Investigations) | 1 | 2
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 2 | 0
HYPERTENSION (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights